CLINICAL TRIAL: NCT06585306
Title: Study on the Safety of High-flow Nasal Oxygen Therapy With Different Flow Rates in Obese Patients Undergoing Sedative Gastroscopy
Brief Title: High-flow Nasal Oxygen Therapy in Obese Patients Undergoing Sedative Gastroscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: XiaoLiang Wang (Other)
Responsible Party: Sponsor-Investigator, XiaoLiang Wang, Chief physician of the Department of Anesthesiology, Perioperative and Pain Medicine, Nanjing First Hospital, Nanjing Medical University, Nanjing, China, Nanjing First Hospital, Nanjing Medical University
Organization: Nanjing First Hospital, Nanjing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY20240419-07
Record Dates: First submitted 2024-05-14; First posted 2024-09-05 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-09

CONDITIONS: Hypoxia; Obesity; Gastrostomy
Keywords: Obese patients; sedative gastroscopy; HFNC
MeSH Terms: conditions — Hypoxia; Obesity | interventions — Intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HFNC30L/min (Experimental): patients pre-oxygenation with pure oxygen at 30L/min for 1 minute, followed by sedation with slightly slow but steady breathing, disappearance of eyelash reflex, and continued oxygen flow at 30 L/min
  Interventions: Behavioral: jaw lift, increasing oxygen flow, mask ventilation, intubation
- HFNC50L/min (Experimental): patients pre-oxygenation with pure oxygen at 30L/min for 1 minute, followed by sedation with slightly slow but steady breathing, adjustment of oxygen flow to 50L/min after disappearance of eyelash reflex.
  Interventions: Behavioral: jaw lift, increasing oxygen flow, mask ventilation, intubation
- HFNC70L/min (Experimental): patients pre-oxygenation with pure oxygen at 30L/min for 1 minute, followed by sedation with slightly slow but steady breathing, adjustment of oxygen flow to 70L/min after disappearance of eyelash reflex.
  Interventions: Behavioral: jaw lift, increasing oxygen flow, mask ventilation, intubation

INTERVENTIONS:
Behavioral: jaw lift, increasing oxygen flow, mask ventilation, intubation — When patients develop hypoxemia, the above interventions are sequentially employed to improve their oxygenation status.

SUMMARY:
Obese patients often have fat accumulation in the head and neck, increased soft tissue in the oropharynx, decreased lung compliance, decreased lung volume and residual volume, and some obese patients also suffer from obstructive sleep apnea. Therefore, obese patients may experience hypoxemia during sedative gastroscopy. High-flow nasal cannula oxygen therapy (HFNC) can provide patients with high-flow (20-70 L/min) and adjustable oxygen concentration (21%-100%) through a special nasal prong catheter. It has the function of warming and humidifying the air, relieving pressure on the nasal mucosa, maintaining airway patency and moisture, reducing the risk of nasal bleeding. In addition, HFNC can generate positive airway pressure (3-7 cmH2O), increase end-expiratory volume, help with alveolar recruitment, prevent atelectasis, and reduce shunts. The flow rate of HFNC is positively correlated with the nasopharyngeal pressure. At a flow rate of 50 L/min, the nasopharyngeal pressure can exceed 3 cmH2O. Obese patients are prone to upper airway obstruction under sedation or anesthesia. The use of HFNC at 70 L/min perioperatively can reduce hypoxemia in patients, but discomfort in the nasopharynx may occur at this flow rate. The optimal flow rate for clinical use of HFNC has not been established. Meta-analysis shows that when the oxygen flow rate during painless esophagogastroduodenoscopy is greater than 30 L/min, it can significantly reduce the incidence of hypoxemia in patients. Therefore, for obese patients undergoing painless esophagogastroduodenoscopy, the investigators propose using HFNC at three different flow rates: 30 L/min, 50 L/min, and 70 L/min, to provide guidance on the optimal flow rate for clinical use of HFNC.

DETAILED DESCRIPTION:
Gastroscopy is a common method for screening and diagnosing digestive diseases, with approximately 23 million cases performed in China annually. However, this invasive procedure can cause patients to experience pain, nausea, vomiting, and coughing. With the advancement of comfortable medical technology, more patients are opting for painless gastroscopy, which offers higher comfort and satisfaction levels for patients and facilitates the operation for endoscopists.

During sedative gastroscopy, nasal cannula oxygen therapy is commonly used to maintain oxygen levels, with oxygen flow rates typically ranging from 2-6L/min. The most common complication during the procedure is hypoxia. For obese patients, the risk of hypoxemia is increased due to fat accumulation in the head and neck, increased soft tissue in the oropharynx, decreased lung compliance and volumes, and potential obstructive sleep apnea. Therefore, appropriate oxygen therapy is crucial in preventing complications in obese patients during gastroscopy.

High-flow nasal cannula oxygen therapy (HFNC) is a new ventilation method that provides patients with high-flow oxygen (20-70L/min) through a special nasal cannula, with adjustable oxygen concentration (21%-100%) and warming and humidifying functionalities. HFNC can alleviate mucosal ciliary pressure, maintain airway patency and moisture, reduce the risk of nasal bleeding, and generate positive airway pressure, aiding in alveolar recruitment and preventing atelectasis.

Studies have shown that HFNC can reduce the occurrence of hypoxia during painless gastroscopy compared to standard oxygen therapy. The positive airway pressure provided by HFNC is crucial in reducing upper airway obstruction and improving ventilation. The optimal flow rate for HFNC in obese patients undergoing gastroscopy remains unclear, but starting at 30L/min has shown benefits in reducing the risk of hypoxemia without significant discomfort.

Therefore, the investigators propose to investigate the effects of HFNC at flow rates of 30L/min, 50L/min, and 70L/min during painless gastroscopy in obese patients to determine the optimal flow rate that minimizes the risk of hypoxemia without causing discomfort.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing sedative gastroscopy
2. Aged over 18.
3. ASA classification I-III
4. Interincisal distance >6.5cm, no micrognathia, limited mouth opening and limited cervical spine movement
5. Compliance with ethics, patient willing to participate in the trial, signed informed consent form

Exclusion Criteria:

1. Contraindications for endoscopic procedures or patients refusing sedation/anesthesia.
2. Patients with allergies to propofol, eggs, soybeans, or milk.
3. Patients with gastrointestinal obstruction and gastric emptying disorders.
4. Patients with acute pharyngitis, tonsillitis, and upper respiratory tract infections.

5: Patients with acute exacerbations of respiratory diseases such as asthma, bronchitis, and COPD. 6. Patients with acute arrhythmias and severe heart disease (congenital, valvular disease). 7. Patients requiring replacement therapy for severe liver or kidney dysfunction.

8. Patients with severe mental illnesses requiring medication to control symptoms.

9. Patients with moderate to severe anemia, coagulation disorders, and hematological diseases. 10. Patients with severe nasal congestion caused by nasal cavity lesions. 11. Pregnant and lactating patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 864 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
incidence of hypoxia | 6 mintues before gastroscopy completion
  75% ≤ SpO2 < 90% for <60 second

SECONDARY OUTCOMES:
incidences of subclinical respiratory depression and severe hypoxia | 6 mintues before gastroscopy completion
  (90% ≤ SpO2 < 95%) and (SpO2 < 75% for any duration or 75% ≤ SpO2 < 90% for ≥60 second)
adverse event | 6 mintues before gastroscopy completion
  vomit
airway obstruction | 6 mintues before gastroscopy completion
  Patients had glossoptosis, excessive oropharynx secretion, laryngeal spasm, or bronchospasm
paradoxical response | 6 mintues before gastroscopy completion
  Patients displayed unpredictable movement, overexcitement, and delirium after sedation with propofol
airway intervention | 6 mintues before gastroscopy completion
  jaw lift, increase the flow of oxygen,mask ventilation,Intubation

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoliang Wang, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No